CLINICAL TRIAL: NCT01425333
Title: The Impact of Surgical Treatment of Ovarian Endometriomas on Ovarian Reserve: a Randomised Controlled Trial of Laparoscopic Ovarian Cystectomy Versus Cyst Ablation - a Pilot Study
Brief Title: The Impact of Surgical Treatment of Endometriomas on Ovarian Reserve
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saad Amer (Other)
Collaborators: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Sponsor-Investigator, Saad Amer, Associate Professor in Gynaecology, University Hospitals of Derby and Burton NHS Foundation Trust
Organization: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R&D: DHRD/2010/089
Record Dates: First submitted 2011-08-25; First posted 2011-08-30 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Endometriosis
Keywords: Ovarian endometriomas; Laparoscopy; Cystectomy; Ablation
MeSH Terms: conditions — Endometriosis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cystectomy (Active Comparator): Patients undergoing cystectomy for ovarian endometrioma
  Interventions: Procedure: Surgery for ovarian endometrioma
- Ablation (Active Comparator): Patients undergoing ablation for ovarian endometrioma
  Interventions: Procedure: Surgery for ovarian endometrioma

INTERVENTIONS:
Procedure: Surgery for ovarian endometrioma — Patients undergoing surgery for ovarian endometrioma
  Other Names: Patients undergoing cystectomy for ovarian endometrioma
  Arms: Cystectomy
Procedure: Surgery for ovarian endometrioma — Patients undergoing surgery for ovarian endometrioma
  Other Names: Patients undergoing cystectomy for ovarian endometrioma
  Arms: Ablation

SUMMARY:
The aim of this study is to assess which of two commonly used surgical procedures in the treatment of ovarian cysts called endometriomas (cutting out of the cyst - "cystectomy", or draining it and cauterising it's inner lining - "ablation") causes the least damage to the ovary and is therefore best at maintaining the future fertility potential of a patient.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing laparoscopic surgery for treatment of unilateral endometriomas measuring ≥ 3cm and ≤ 8cm in diameter

Exclusion Criteria:

* Patients who have received oestrogen suppressing drugs (e.g. oral contraceptive pills, GnRHa) during the previous six months
* Patients who have previously undergone surgical treatment of endometriomas
* Patients with bilateral endometriomas
* Patients with endometriomas of less than 3cm in size or more than 8cm in size
* Pre-surgical evidence of reduced ovarian reserve
* Pregnant patients
* Patients unable to give informed consent e.g. patients with mental incapacity

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-08 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Anti-Mullerian Hormone (AMH) | 6 months post-operatively
  Change in anti-mullerian hormone level after surgery (at one week, three months and six months)

SECONDARY OUTCOMES:
Follicle Stimulating Hormone (FSH) | 6 months
  Change in follicle stimulating hormone levels after surgery (at one week, three months and six months)
Antral Follicle Count (AFC) | 3 months
  Change in AFC after surgery (at three months)

CONTACTS AND LOCATIONS:
Overall Officials: Saad Amer, MD, MRCOG, Principal Investigator — University of Nottingham and Derby Hospitals NHS foundation Trust
Locations (1):
- Royal Derby Hospital, Derby, United Kingdom